CLINICAL TRIAL: NCT06270823
Title: Making Elective Caesarean Safer for Infant's Lungs by Reducing Respiratory Distress Using Knee-chest-flexion: a Randomized Controlled Trial
Brief Title: Reducing Respiratory Distress After Elective Caesarean Birth Through Knee-chest-flexion: a Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kilimanjaro Clinical Research Institute (Other)
Collaborators: Leiden University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NIMR/HQ/R.8a/Vol.IX/4331
Record Dates: First submitted 2024-02-14; First posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Transient Tachypnea of the Newborn
Keywords: planned caesarean birth
MeSH Terms: conditions — Transient Tachypnea of the Newborn

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- interventional arm (Experimental): As soon as the infant is out of the uterus a Knee-to-chest flexion (KCF) maneuver is performed for 30 seconds while the infant remains attached to the cord. When applying KCF, we essentially bring the newborn back into the fetal position, flexing the knees to the chest. This is similar to the holding position applied for performing lumbar puncture in neonates. Except for KCF, the infant will receive normal routine care and there are no co-interventions.
  Interventions: Procedure: Knee-to-chest-flexion manoeuvre
- control (No Intervention): As soon as the infant is out of the uterus normal routine care is given

INTERVENTIONS:
Procedure: Knee-to-chest-flexion manoeuvre — The obstetrician will place one hand at the neck and shoulder of the baby and gently bend the infant into dorsiflexion while with the other hand bending the hips and knees against the abdomen and chest (squatting into fetal position). This holding position will be continued for 30 seconds, while compression of the umbilical cord is avoided to maintain an undisturbed umbilical circulation to and from the infant during KCF.
  Arms: interventional arm

SUMMARY:
Planned caesarean birth is a risk factor for the development of neonatal respiratory distress commonly known as transient tachypnoea of the newborn. This is due to the absence of labor physiology which facilitates the clearance of fetal lung fluid. We hypothesized that by mimicking flexion induced by uterine contractions by manually performing knee-to-chest flexion directly at birth to achieve expulsion of excess lung liquid, we could reduce the incidence of respiratory distress in term children born by planned CS.

The goal of this clinical trial is to test whether performing a knee-to-chest flexion maneuver directly after elective caesarean section will decrease the incidence of respiratory distress in term infants when compared to the standard care

DETAILED DESCRIPTION:
One of the major risk factors for term/near-term infants to develop respiratory distress (RD) is when they are born by elective caesarean section (CS). While this form of RD, commonly diagnosed as transient tachypnea of the newborn (TTN), is considered to be self-limiting, the severity of RD often leads to unexpected admission to the pediatric ward for respiratory support. TTN has also been associated and asthma, bronchiolitis, and other wheezing syndromes later in life. In low- and middle-income settings, where neonatal intensive care resources are limited, a considerable proportion of babies in need of respiratory support do not survive.

There is now strong physiological evidence that RD after elective cesarean section is caused by this greater volume of airway liquid present at birth, which is due to the absence of labor. During labor, uterine contractions contribute to the flexion of the fetus which increases abdominal and transpulmonary pressure. This elevates the diaphragm, resulting in lung liquid loss via nose and mouth. Flexion induced by uterine contractions could be mimicked by manually performing knee-to-chest flexion directly at birth, to achieve expulsion of excess lung liquid. When applying KCF, we essentially bring the newborn back into fetal position, similar to the holding position applied for performing lumbar puncture in neonates.

If this simple intervention has shown to improve neonatal outcome in the clinical setting, KCF will undoubtedly be an extremely cost-effective health care innovation. The maneuver is easy-to-teach to any clinician performing cesarean section. KCF will be performed conform standard gentle care and is likely to be entirely harmless. These advantages (easy-to-teach, no cost, no harm) are relevant across all settings, but may be particularly appealing in low-income settings, where neonatal follow-up and access to neonatal intensive care are often either impossible or limited. It is therefore of outmost importance to test this intervention in a larger institution adapted to performing high-quality clinical research in a low- or middle-income country.

We now hypothesize that performing a knee-to-chest flexion performed directly after birth will reduce the incidence of respiratory distress in term children born by elective caesarean section.

Objective: To test whether performing a knee-to-chest flexion (KCF) manoeuvre directly after elective CS will decrease the incidence of respiratory distress in term infants when compared to standard care.

Study design: Single-center randomized controlled trial Study population: Infants born by elective CS, 37-42 weeks gestational age. Simple randomization will be done to assign participants in either an interventional group or a control group Intervention: As soon as the infant is out of the uterus a KCF is performed for 30 seconds while the infant remains attached to the cord. Except for KCF, the infant will receive normal routine care and there are no co-interventions.

Control: As soon as the infant is out of the uterus normal routine care is given.

Study parameters: The primary outcome is the occurrence of respiratory distress

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

In the group of term infants born after elective caesarean there is a 7% risk for respiratory distress, of which 10% is complicated by PPHN. Although KCF is a new intervention performed directly after birth for 30 seconds, the technique used is similar to the way infants are held and positioned during a lumbar puncture. As the infants in this study population are in good condition before birth and would otherwise also have been exposed to large intrathoracic pressures generated by uterine contractions during labor, we expect that there is no added risk when the maneuver is performed gently and with care. We recently demonstrated that performing KCF directly after birth is feasible and safe after elective CS. As the percentages of elective CS are increasing worldwide both in developing and developed countries, there is a large potential to reduce morbidity, admissions at NICU and pediatric wards, and healthcare costs in this group of infants.

ELIGIBILITY:
Inclusion Criteria:

* Infants born by planned CS, 37-42 weeks gestational age

Exclusion Criteria:

* infants with significant congenital malformations influencing cardiopulmonary transition
* infants whose mother has gestational diabetes, pre-eclampsia, eclampsia
* infants where immediate cord clamping is needed due to resuscitation of the baby or mother
* when spontaneous contractions before the cesarean section is done.
* KCF will not be done to infants who will start breathing instantly after being extracted from the uterus so as not to interfere with their breathing efforts

Max Age: 30 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 562 (Estimated)
Dates: Start 2024-02-14 (Actual); Primary Completion 2025-02-14 (Estimated); Study Completion 2025-02-14 (Estimated)

PRIMARY OUTCOMES:
respiratory distress | 24 hours
  newborns who have any signs of respiratory distress such as tachypnoea, nasal flaring, chest indrawing, grunting, cyanosis

SECONDARY OUTCOMES:
adverse outcome of knee-to-chest flexion maneuver | 24hours
  any signs of adverse outcomes from knee to chest flexion maneuver such as Hematoma on extremities, abdomen, or chest within 24 hours after birth

CONTACTS AND LOCATIONS:
Overall Officials: Bariki Mchome, PhD, Principal Investigator — Kilimanjaro Christian Medical Centre; Blandina T Mmbaga, PhD, Principal Investigator — Kilimanjaro Clinical Research Institute; Febronia L Shirima, MD, Principal Investigator — Kilimanjaro Clinical Research Institute
Locations (1):
- Kilimanjaro Christian Medical Centre, Moshi, Kilimanjaro, Tanzania

IPD SHARING:
Plan to Share IPD: Yes
Individual Participant Data that underlies results in a publication will be shared
Supporting Information: Study Protocol
Time Frame: Beginning 3 months following publication. No end date
Access Criteria: Researchers who provide a methodologically sound proposal. Proposals should be directed to A.B.te_Pas@lumc.nl. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Shirima FL, Keus A, Mchome B, Mangi G, Davies I, van den Akker T, Mmbaga BT, Hooper SB, Te Pas AB. The effectiveness of knee-chest-flexion maneuver in reducing respiratory distress in elective cesarean section newborns: protocol for a randomized controlled trial. Contemp Clin Trials. 2025 Sep;156:108006. doi: 10.1016/j.cct.2025.108006. Epub 2025 Jul 11. PMID 40653309